CLINICAL TRIAL: NCT05638087
Title: Dexamethasone as a Novel Treatment for Obstructive Sleep Apnea in Children
Brief Title: Dexamethasone Treatment for OSA in Children
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Indra Narang, Senior Associate Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000079288
Record Dates: First submitted 2022-11-02; First posted 2022-12-06 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Dexamethasone; Corticosteroid
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone Treatment (Experimental): Oral Dexamethasone treatment
  Interventions: Drug: Dexamethasone
- Placebo Treatment (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone Oral Suspension
  Arms: Dexamethasone Treatment
Drug: Placebo Control — Placebo Oral Mix
  Arms: Placebo Treatment

SUMMARY:
This is a double-blinded clinical trial of children diagnosed with moderate to severe obstructive sleep apnea (OSA) on a baseline polysomnogram (PSG). Participants will receive a 3-day course of dexamethasone, an oral steroid, or placebo control and undergo two PSGs to assess the efficacy of dexamethasone, as a treatment to manage the severity and symptoms in children with moderate to severe OSA.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common sleep-related breathing disorder affecting neonates to adolescents characterized by intermittent partial and complete upper airway obstruction leading to apneas.

The first line of treatment for OSA in young children is an adenotonsillectomy (AT). However, there are long surgical wait times for ATs, up to 3-6 months after a baseline polysomnogram(PSG). This leaves many children untreated, leading to a higher risk of learning deficits and long-term health effects.

Oral corticosteroids have long been used to treat airway inflammation and reduce inflammation of adenoid and tonsil tissue in-vitro. However, there is a lack of knowledge of oral steroids' efficacy in managing OSA. Additionally, the role of the nasal epithelium and the mechanism of action of dexamethasone role at a molecular level is unknown.

The primary objective is to evaluate the efficacy of Dexamethasone in reducing the severity and symptoms of moderate to severe OSA in children in this proof-of-concept exploratory trial.

Participants will be screened by their baseline PSG, followed by 3 study visits conducted at SickKids. Participants will receive a 3-day course of oral dexamethasone or placebo at their first baseline study visit. During baseline, participants will undergo an otolaryngology assessment, a nasal brushing, and questionnaires. Participants will return 2 to 4 weeks after the intervention to the Hospital for Sick Children for a follow-up study visit which includes a repeat PSG, otolaryngology assessment and questionnaires. If no AT is performed within 6 months, participants will return for a third study visit for a repeat PSG, otolaryngology assessment and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Polysomnogram diagnosed with moderate to severe Obstructive sleep apnea (OAHI >5 events/hour)
* Aged 2-10 years
* Presence of adenotonsillar hypertrophy
* Ability to take oral medication and be willing to adhere to the dosing regimen
* Informed consent provided in accordance with institutional policies

Exclusion Criteria:

* Previous adenotonsillectomy
* Presence of symptoms of an upper respiratory tract infection
* Co-existing central sleep apnea
* Hypertension
* Prior or current evidence for abnormal glucose tolerance
* Contraindication for dexamethasone or components of dexamethasone oral suspension,
* Treatment with nasal or systemic corticosteroids within 4 weeks prior to the intervention
* OSA with associated oxygen desaturations <90% for 2 continuous minutes
* Need for non-invasive ventilation long-term due to underlying disease
* Current systemic fungal infections
* Patients with clinically relevant varicella exposure

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-07-21 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Obstructive apnea-hypopnea index | Baseline and 2-4 weeks
  Change in obstructive apnea-hypopnea index from baseline.
  The paediatric OSA severity scoring criteria will be used for all participants. Mild OSA is defined as OAHI ≥1 to <5 events/hr; moderate OSA is defined as OAHI ≥5 to <10 events/hr; and severe OSA is defined as OAHI ≥10 events/hr

SECONDARY OUTCOMES:
Change in scores from baseline of the Child Sleep Habits Questionnaire (CSHQ) total score | Baseline and 2-4 weeks
  Total CSHQ score of 41 has been reported to be a sensitive clinical cut-off point for detecting possible sleep problems
Change in scores from baseline of the Strengths and Difficulties Questionnaire (SDQ) | Baseline and 2-4 weeks
  The SDQ is a validated parent-reported behavioural screening questionnaire and is used to assess children's mental health. The total difficulties score ranges from 0 to 40, a higher score indicates higher difficulties.
Change in scores from baseline of the Obstructive Sleep Apnea-18 Quality of Life (OSA-18 QoL) Survey. | Baseline and 2-4 weeks
  The OSA-18 QoL survey is a validated 18-item quality of life measure for children with sleep-disordered breathing (SDB) for children 2-18. Higher total scores indicate more impact on QoL - minor impact (scores below 60), moderate impact (scores between 60 and 80) and major impact (scores above 80).
Soft tissue size (Adenoids, Tonsils & Turbinates) | Baseline and 2-4 weeks
  Change in soft tissue size (adenoids, tonsils and turbinates) from baseline
Cytokine levels of Interleukin-8(IL-8), Interleukin-1b(IL1b), and Tumor Necrosis Factor a (TNFa) at baseline | At baseline
  Inflammatory markers will be measured in basal media of cells cultured from nasal brushing by ELISA
Inflammatory gene expression of Interleukin-8, Interleukin-1b, Nuclear factor kappa-B (NF-kB) and Tumor Necrosis Factor a (TNFa) | At baseline
  Cells from nasal brushing will be cultured and harvested for RNA to study gene expression.
Participant recruitment rate | From study start to completion; up to 6 months
  Feasibility determined by participant recruitment rate
Participant retention rate | From study start to completion; up to 6 months
  Feasibility determined by participant retention rate
Participant adherence rate | From study start to completion; up to 6 months
  Feasibility determined by participant adherence rate
Adverse events | From study start to completion; up to 6 months
  Safety determined by number and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Indra Narang, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No